CLINICAL TRIAL: NCT06790966
Title: A Phase 3 Open-Label, Randomized Study of PDS0101 and Pembrolizumab vs Pembrolizumab Alone in First-Line Treatment of Unresectable Recurrent and/or Metastatic HPV16+ Head and Neck Squamous Cell Carcinoma
Brief Title: Phase 3 Study of PDS0101 and Pembrolizumab in HPV16+ Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Acronym: VERSATILE-003
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PDS Biotechnology Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDS0101-HNC-301
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Head and Neck Cancer; Metastatic Head and Neck Cancer; HPV Positive Oropharyngeal Squamous Cell Carcinoma; Neoplasms, Head and Neck; Unresectable Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck cancer; Head and neck neoplasms; Neoplasms, squamous cell; Squamous cell carcinoma of the head and neck; Head and neck squamous cell carcinoma; Recurrent Head and Neck cancer; Metastatic Head and Neck Cancer; Immuno-oncology therapy; Human papillomavirus-16; Cancer Vaccines; HNSCC; Oropharyngeal squamous cell carcinoma; HPV; Programmed cell death ligand 1; PD-L1; Immune checkpoint inhibitor; Immune checkpoint inhibitors; Immunotherapy; Squamous cell cancer; Pembrolizumab; Antineoplastic Agents, Immunological
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a Phase 3 open-label, active-control, 2:1 randomized study with parallel assignment of PDS0101 plus pembrolizumab (referred to as 'the investigational arm') vs pembrolizumab alone (referred to as 'the control arm')
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Experimental): PDS0101 + Pembrolizumab
  Interventions: Combination Product: Combination Treatment of PDS0101 and Pembrolizumab
- Control Arm (Active Comparator): Pembrolizumab
  Interventions: Drug: Pembrolizumab Monotherapy

INTERVENTIONS:
Combination Product: Combination Treatment of PDS0101 and Pembrolizumab — * Pembrolizumab (IV) every 3 weeks for up to 35 Cycles
  * PDS0101 (SC) during Cycles 1, 2, 3, 4, and 12
  Other Names: Versamune HPV; KEYTRUDA
  Arms: Interventional Arm
Drug: Pembrolizumab Monotherapy — Pembrolizumab (IV) every 3 weeks for up to 35 cycles.
  Other Names: KEYTRUDA
  Arms: Control Arm

SUMMARY:
This is a global, multi-center, Phase 3 study that is randomized 2:1, controlled, and open label to evaluate PDS0101 (Versamune + HPVMix) in combination with pembrolizumab vs. pembrolizumab monotherapy as first-line treatment in patients with unresectable recurrent or metastatic HPV16-positive HNSCC expressing programmed cell death ligand-1 (PD-L1) with combined positive score (CPS) ≥1.

DETAILED DESCRIPTION:
PDS0101 is a T cell activating immunotherapy designed to induce HPV-specific CD8 and CD4 T cells. A Phase 2 study has shown promising signs of safety and efficacy when PDS0101 is combined with pembrolizumab in patients with HPV16-positive R/M HNSCC with CPS ≥1, which is the population for this study.

The primary objective of this study is to compare the effect of the combination of PDS0101 plus pembrolizumab vs. pembrolizumab monotherapy on overall survival. Secondary objectives for this study include comparison of effects on objective response rate (ORR), disease control rate (DCR), duration of response (DOR), and progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Subject (or legally acceptable representative, if applicable) provides written informed consent for the study.
2. Subject is ≥18 years of age on the day of signing the informed consent.
3. Have a history of histologically- or cytologically-confirmed diagnosis of recurrent and/or metastatic squamous cell cancer of the head and neck (HNSCC) with:

   1. Eligible primary tumor location of oropharynx, oral cavity, hypopharynx, or larynx.
   2. HPV16 tumor positivity (central testing).
   3. Tumor PD-L1 expression defined as a CPS ≥ 1 using the FDA- approved pembrolizumab (KEYTRUDA®) assay (local testing).
   4. No prior systemic anticancer therapy administered in the incurable recurrent or metastatic setting. Systemic therapy which was completed more than 6 months prior to randomization, if given as part of multimodal treatment for locally advanced disease, is allowed.
4. Have measurable disease based on RECIST 1.1 as determined by the site and confirmed by BICR. As a guidance to the site investigators, tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
5. Subject has adequate organ function defined by the following parameters (all specimens must be collected within 15 days prior to randomization):

   * Hematological: Absolute neutrophil count (ANC) ≥1500/μL, Platelets ≥100,000/μL; Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L;
   * Renal: Estimated glomerular filtration rate ≥30 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
   * Hepatic: Total bilirubin ≤1.5 × ULN or direct bilirubin ≤ULN for subjects with total bilirubin levels >1.5 × ULN, Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.5 ULN (if approved by Medical Monitor, ≤5 × ULN for subjects with liver metastases; AST and ALT >5 to 20 x ULN may be included if asymptomatic).
   * Coagulation: INR, prothrombin time (PT) ≤1.5 × ULN; if subject is receiving anticoagulant therapy, INR or PT- should be within therapeutic range of anticoagulant.
6. For female subjects defined as women of childbearing potential (WOCBP), a negative urine pregnancy test must be obtained during screening. If the urine test cannot be confirmed as negative, a serum pregnancy test will be required. Women who are surgically sterile or at least 2 years postmenopausal do not require pregnancy testing.
7. Male subjects of childbearing potential must agree to use a condom as an effective method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

1. Primary tumor location of nasopharynx (any histology).
2. If the urine pregnancy test is positive. If the urine test cannot be confirmed as negative, a serum pregnancy test will be required.
3. Has received prior therapy with HPV-specific immunotherapy including therapeutic cancer vaccines and cellular immunotherapy. Note: subjects who have received prophylactic HPV vaccines are eligible for enrollment.
4. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD- L2 agent or with an agent directed to another stimulatory or co- inhibitory T cell receptor including but not limited to CTLA-4, OX40, CD137.
5. Has had major surgery, including surgical resection of tumor, within 30 days prior to randomization, and has not fully recovered as assessed by the investigator.
6. Has received radiotherapy prior to randomization outside of the following minimum washout periods, and has not fully recovered as assessed by the investigator:

   * Fractionated radiotherapy, 2 weeks
   * Stereotactic radiosurgery, 1 week
   * Palliative radiation therapy, 1 week
7. Has received a live vaccine within 30 days prior to randomization.

   Examples of live vaccines include, but are not limited to, the following:

   measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed-virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist ® ) or live attenuated vaccines are not allowed within 30 days prior to randomization.
8. Has received immunomodulatory or immunosuppressive agents (e.g., interferons (IFNs), tumor necrosis factor, interleukins, immunoglobulins or other biological response modifiers (granulocyte colony-stimulating factor [GCSF] or granulocyte macrophage stimulating factor [GMCSF]) within 30 days prior to randomization.
9. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 30 days prior to randomization. Note: Subjects who entered the follow-up phase of an investigational study may participate as long as it is permitted in that study consent and has been 30 days after the last dose of the previous investigational agent.
10. Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years. Note: Subjects who have had a transplant greater than 5 years ago are eligible as long as there are no symptoms of graft- versus-host disease [GVHD].
11. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (I a dose exceeding 10 mg daily of prednisone equivalent). Note: Current or recent use of intranasal, intra-articular, and topical steroids are allowed for symptom management are clinically indicated.
12. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Subjects with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ, superficial [non- infiltrated] bladder tumors) or other malignant tumors that have undergone potentially curative therapy are eligible for enrollment.
13. Has known carcinomatous meningitis and/or active central nervous system (CNS) metastases as defined by new brain metastases or progressive brain metastases that have not been subjected to CNS-directed therapy since documented progression. Note: Subjects with previously treated brain metastases are eligible if all the following criteria are met:

    1. radiologically stable, i.e., without evidence of progression for at least 30 days by repeat imaging (note that repeat imaging should be performed during study screening),
    2. neurologically stable, and
    3. without requirement of steroid treatment for at least 14 days prior to randomization.
14. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered systemic treatment and is allowed.
15. Has a history of interstitial lung disease or has current pneumonitis. Note: Subjects with a history of radiation pneumonitis who are fully recovered are eligible.
16. Has an active infection requiring systemic therapy (e.g., IV or oral anti-infective).
17. Has known human immunodeficiency virus (HIV) and CD4 count < 350 cells/μL and/or a history of an AIDS-defining opportunistic infection within the past 12 months. Note: Subjects who are on stable antiretroviral therapy for at least 30 days and have an HIV viral load less than 400 copies/mL and who do not meet the above exclusion criterion may be enrolled.
18. Has a history of hepatitis B (HBV) infection or known to be positive for HBV antigen (HbsAg)/HBV virus DNA.
19. Has active hepatitis C defined by a known positive C Ab result and known quantitative HCV RNA results greater than the lower limits of detection of the assay. Note: Subjects with a history of HCV infection who have completed curative antiviral treatment and have HCV viral load below the limit of quantification may be enrolled.
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study.
22. Is breastfeeding within the projected duration of the study, starting with the screening visit through 120 days after the last dose of any study treatment.
23. Has had an allogenic tissue/solid organ transplant.
24. Female subjects defined as WOCBP unwilling or unable to use highly effective contraception method(s) for the duration of the study:

    1. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation.
    2. Progestogen-only hormonal contraception
    3. Intrauterine device
    4. Intrauterine hormone-releasing system
    5. Bilateral tubal occlusion
    6. Vasectomized partner is a highly effective birth control method provided that the partner is the sole sexual partner of the women of childbearing potential (WOCBP) trial participant and that the vasectomized partner has received medical assessment of surgical success.
25. History of allergic or hypersensitivity reactions (≥Grade 3) to pembrolizumab, PDS0101, or their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 48 months
  OS is defined as the time from randomization until death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 27 months
  ORR is defined as the percentage of subjects with an objective response: a complete response (CR) or partial response (PR) using RECIST 1.1 criteria as assessed by BICR.
Disease Control Rate (DCR) | Up to 27 months
  DCR is defined as the percentage of subjects with an objective response of CR, PR, or stable disease (SD, at least 6 weeks after first dose) using RECIST 1.1 criteria as assessed by BICR.
Duration of Response (DOR) | Up to 27 months
  DOR is defined as the time from initial response to disease progression or death as determined by using RECIST 1.1 criteria as assessed by BICR.
Progression-Free Survival (PFS) | Up to 27 months
  PFS is defined as the time from randomization until disease progression or death from any cause, whichever occurs first. PFS will be based on RECIST 1.1 as assessed by BICR.

OTHER OUTCOMES:
Safety | Up to 48 months
  Adverse events (AEs), serious adverse events (SAEs), and discontinuation due to AEs.
Progression-Free Survival 2 (PFS2) | Up to 48 months
  Defined as the time from randomization to second disease progression after initiation of an anti-cancer therapy following discontinuation of study treatments, or death from any cause, whichever comes first.
European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3L) | Up to 48 months
  Change from baseline and time to deterioration.
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQC30) | Up to 48 months
  Change from baseline and time to deterioration.
EORTC Quality of Life - Head and Neck Cancer Module (QLQH&N35) | Up to 48 months
  Change from baseline and time to deterioration.
ORR | Up to 27 months
  By RECIST 1.1 investigator assessment.
Immune-related (ir)ORR | Up to 27 months
  By irRECIST.
DCR | Up to 27 months
  By RECIST 1.1 investigator assessment.
DOR | Up to 27 months
  By RECIST 1.1 investigator assessment.
PFS | Up to 27 months
  By RECIST 1.1 investigator assessment.
Immune-related (ir)DCR | Up to 27 months
  By irRECIST.
Immune-related (ir)DOR | Up to 27 months
  By irRECIST.
Immune-related (ir)PFS | Up to 27 months
  By irRECIST.

CONTACTS AND LOCATIONS:
Overall Officials: David Schaaf, MD, Study Director — PDS Biotechnology Corporation
Locations (28):
- United States (28):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Marin Cancer Care, Greenbrae, California
  - University of California, Orange, Orange, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Florida Cancer Affiliates - Ocala Oncology, Ocala, Florida
  - SCRI - Florida Cancer Specialists, Orlando, Florida
  - Emory University - Winship Cancer Institute (WCI), Atlanta, Georgia
  - University of Kansas, Westwood, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - The Ohio State University- James Cancer Hospital, Columbus, Ohio
  - Penn State Health, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Texas Oncology, Austin, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Texas Oncology-Northeast Texas, Tyler, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - West Virginia University Cancer Center, Morgantown, West Virginia